CLINICAL TRIAL: NCT03633825
Title: Randomized Controlled Trial of an Online Machine Learning-Driven Risk Assessment and Intervention Platform for Increasing the Use of Crisis Services
Brief Title: Brief Online Help-seeking Barrier Reduction Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Adam Jaroszewski, Principal Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB17-1303
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Results first posted 2019-04-17 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Crisis Intervention; Suicide and Depression
Keywords: suicide; mental health crisis; crisis referrals; help-seeking; risk assessment; treatment barrier
MeSH Terms: conditions — Suicide; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Brief help-seeking barrier reduction intervention

INTERVENTIONS:
Behavioral: Brief help-seeking barrier reduction intervention — The BRI was designed to overcome common concerns and misconceptions (i.e., barriers) related to using crisis services. It works by first asking the user about what potential barriers may keep them from using the crisis service referrals, and then, based on the user's response, by providing information intended to help the user overcome the potential barrier(s) they selected. By exploring the menu of barriers, users could read brief messages designed to dispel common misconceptions or concerns related to each barrier. For example, a common concern among Koko users was that calls to lifelines invariably result in visits by the police or other emergency services. Users who feared this possibility could tap on the associated button and learn that active rescues such as these are extremely rare, and occur in less than one percent of all cases. Whenever possible, we used language throughout the intervention to help validate the experiences of the users.
  Arms: Intervention

SUMMARY:
Objective: Mental illness is a leading cause of disease burden; however, many barriers prevent people from seeking mental health services. Technological innovations may improve the ability to reach under-served populations by overcoming many existing barriers. The investigators evaluated a brief, automated risk assessment and intervention platform designed to increase the use of crisis resources provided to individuals who were online and in crisis. Hypothesis: The investigators hypothesized that individuals assigned to the intervention condition would report using crisis resources at higher rates than individuals in the control condition. Method: Participants, users of the digital mental health app Koko, were randomly assigned to treatment or control conditions upon accessing the app and were included in the study after their posts were identified by machine learning classifiers as signaling a current mental health crisis. Participants in the treatment condition received a brief Barrier Reduction Intervention (BRI) designed to increase the use of crisis service referrals provided on the app. Participants were followed-up several hours later to assess the use of crisis services.

ELIGIBILITY:
Inclusion Criteria:

* Participants identified as experiencing a mental health crisis by a hybrid human-machine computation system evaluating semantic content of posts made on digital platforms.

Exclusion Criteria:

* Participants who were not identified as experiencing a mental health crisis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39450 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaroszewski AC, Morris RR, Nock MK. Randomized controlled trial of an online machine learning-driven risk assessment and intervention platform for increasing the use of crisis services. J Consult Clin Psychol. 2019 Apr;87(4):370-379. doi: 10.1037/ccp0000389. PMID 30883164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 39,450 Koko users who signed up for the service between August 10, 2017 and September 20, 2017. Koko (née Panoply) provides safety services for large online social networks.
Pre-assignment Details: All potential participants (N=39,450) screened for eligibility were considered enrolled. Potential participants were randomized upon accessing the platform, not later when identified as being in-crisis, because we used the platform's extant, AB-testing randomization tool. No other AB-tests were on the platform during the study period.
Groups:
- Control: Control Condition: Users in the control condition experienced the Koko digital platform as usual.
- Intervention: Brief help-seeking barrier reduction intervention: The BRI was designed to overcome common concerns and misconceptions (i.e., barriers) related to using crisis services. It works by first asking the user about what potential barriers may keep them from using the crisis service referrals, and then, based on the user's response, by providing information intended overcome the potential barrier(s) they selected. By exploring various barriers, users could read brief messages designed to dispel common misconceptions/concerns related to each barrier. For example, a previous study among Koko users found that a common concern was that calls to lifelines invariably result in visits by the police. Users who feared this possibility could tap on the associated button and learn that active rescues such as these are extremely rare, and occur in less than one percent of all cases. Whenever possible, we used language throughout the intervention to help validate the experiences of the users.
Period: Enrollment
Arm/Group | Control | Intervention
Started (Randomized and assessed for eligibility.) | 19838 | 19612
Completed | 805 | 775
Not Completed | 19033 | 18837
Not completed — Did not post on network | 5066 | 5080
Not completed — Post not classified as crisis | 13967 | 13757
Period: Allocation
Arm/Group | Control | Intervention
Started (Allocated and received intervention.) | 805 | 775
Completed | 805 | 775
Not Completed | 0 | 0
Period: Follow up
Arm/Group | Control | Intervention
Started | 805 | 775
Completed | 327 | 325
Not Completed | 478 | 450
Not completed — Lost to Follow-up | 478 | 450
Period: Analysis
Arm/Group | Control | Intervention
Started | 327 | 325
Completed | 327 | 325
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Brief help-seeking barrier reduction intervention: The BRI was designed to overcome common concerns and misconceptions (i.e., barriers) related to using crisis services. It works by first asking the user about what potential barriers may keep them from using the crisis service referrals, and then, based on the user's response, by providing information intended overcome the potential barrier(s) they selected. By exploring various barriers, users could read brief messages designed to dispel common misconceptions/concerns related to each barrier. For example, a common concern among Koko users was that calls to lifelines invariably result in visits by the police. Users who feared this possibility could tap on the associated button and learn that active rescues such as these are extremely rare, and occur in less than one percent of all cases. Whenever possible, we used language throughout the intervention to help validate the experiences of the users.
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 805 | 775 | 1580
Age, Continuous [Mean (Standard Deviation); unit: years] — Participant age was not collected. Population: Age was not collected.
Sex: Female, Male [Count of Participants; unit: Participants] — Participant sex was not collected. Population: Sex was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Participant region of enrollment was not collected. Population: Region of Enrollment was not collected.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Use of Crisis-referrals
Description: The number participants indicating at follow-up that they used the crisis resources provided to them (e.g., called the suicide crisis hotline)
Time Frame: 5 hours post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 327 | 325
Participants | 130 | 159
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .02, Chi-squared; Risk Ratio (RR) = 1.23, 95% CI 2-sided [1.03 to 1.46]

2. Secondary Outcome: Number of Participants in the Treatment Versus Control Conditions Reporting Their Experience Using Koko Was "Good"
Description: The number of participants in the treatment versus control conditions reporting that their experience on the Koko digital platform was "good" versus "bad" using a two-option response question.
Time Frame: 5 hours post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 327 | 325
Participants | 250 | 234
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = .19, Chi-squared; Risk Ratio (RR) = 1.2, 95% CI 2-sided [0.91 to 1.59]

ADVERSE EVENTS:
Time Frame: 31 days.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/805 | 0/775
Serious Adverse Events (participants affected / at risk) | 0/805 | 0/775
Other Adverse Events (participants affected / at risk) | 0/805 | 0/775

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT03633825/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT03633825/SAP_000.pdf